CLINICAL TRIAL: NCT01473732
Title: Mechanisms and Treatment of Chronic Allograft Injury (CAI) Due to Calcineurin Inhibitor (CNI) Toxicity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: terminated after 2 patients due to difficulty in enrollment
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Enver Akalin, Prof. Dept of Medicine (Nephrology), Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-05-196
Record Dates: First submitted 2011-11-14; First posted 2011-11-17 (Estimated); Results first posted 2018-09-18 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: Chronic Allograft Injury; Calcineurin Inhibitor Toxicity
Keywords: CNI toxicity; CAI
MeSH Terms: interventions — Everolimus; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Everolimus (Zortress) (Experimental)
  Interventions: Drug: Everolimus; Drug: Mycophenolic acid
- Reduced dose Tacrolimus (Prograf) (Active Comparator)
  Interventions: Drug: Tacrolimus; Drug: Mycophenolic acid

INTERVENTIONS:
Drug: Everolimus — Starting dose 1.5 mg bid, target trough level 6-10 ng/ml.
  Other Names: Zortress
  Arms: Everolimus (Zortress)
Drug: Tacrolimus — Target trough level of Tacrolimus 3-5 ng/ml.
  Other Names: Prograf
  Arms: Reduced dose Tacrolimus (Prograf)
Drug: Mycophenolic acid — Myfortic Min. dose 360 mg bid and Max dose 720 mg bid. Used in both arms. Used for one year.
  Other Names: Myfortic

SUMMARY:
The purpose of this study is to find out how well the current drug regimen (including low Prograf dose and Myfortic, which is usually recommended to prevent any further deterioration in the kidney function) works and how safe it is when compared to a combination of Zortress and Myfortic in patients with chronic kidney injury associated with Prograf or Neoral use.

DETAILED DESCRIPTION:
Specific Aim 1: To investigate allograft and peripheral blood cell gene expression patterns of patients with CAI by using Affymetrix microarrays.

Hypothesis 1: Gene expression patterns of patients with biopsy findings suggesting calcineurin inhibitor (CNI) toxicity without significant tubulointerstitial infiltrates or transplant glomerulopathy might demonstrate upregulation of genes related to tissue injury, fibrosis, and extracellular matrix deposition without upregulation of genes related to alloimmune response, such as, T and/or B lymphocyte activation markers, surface receptors, co-stimulation molecules, adhesion molecules, cytokines, and chemokines comparing to patients with significant tubulointerstitial infiltrates and/or transplant glomerulopathy that might show upregulation of genes related to alloimmune response, such as, T and/or B lymphocyte activation markers, surface receptors, co-stimulation molecules, adhesion molecules, cytokines, and chemokines.

Specific Aim 2: The effect of everolimus (Zortress)/ mycophenolate sodium (EC-MPS, myfortic®) treatment on allograft and peripheral gene expression patterns.

Hypothesis 2: Everolimus (Zortress) and mycophenolate sodium (EC-MPS, myfortic®) treatment attenuates the progression of CAI due to CNI toxicity by downregulating the expression of genes related to fibrosis, such as, transforming growth factor-β, thrombospondin 1, and platelet derived growth factor-C.

Specific Aim 3: To document the clinical outcomes of everolimus (Zortress) and mycophenolate sodium (EC-MPS, myfortic®) in patients with CAI due to CNI toxicity Hypothesis 3: Everolimus (Zortress) and mycophenolate sodium (EC-MPS, myfortic®) can attenuate the progression of CAI due to CNI toxicity and may improve the creatinine clearance.

ELIGIBILITY:
Inclusion Criteria:

All patients with biopsy proven pure chronic allograft injury due to CNI toxicity.

Exclusion Criteria:

1. 24 hour urine protein or spot urine protein/creatinine ratio > 500 mg/day
2. Estimated glomerular filtration rate (eGFR) < 30 ml/min by modification of Diet in Renal Disease( MDRD) or 24 hour urine collection
3. Patients with Donor-specific antibody (DSA) by Luminex (mean fluorescence intensity values > 1,000)
4. Recipients of multiple organ transplants or ABO-incompatible allograft
5. Current panel reactive antibody (PRA) greater than 30 percent
6. Graft loss at randomization
7. Pregnant women
8. Previous history of acute rejection
9. Previous history of allergy or intolerance to Zortress or Myfortic
10. Platelet count less than 100,000
11. White Blood Cell (WBC) less than 3,000
12. Hb less than 9 g/dL or Htc less than 30%
13. Biopsy findings of

    * Chronic antibody mediated rejection
    * Acute rejection
    * Positive C4d staining
    * Interstitial infiltrates more than 25% of the area
    * Transplant glomerulopathy
    * Recurrent or de novo glomerular disease
    * Polyoma nephropathy or positive simian virus 40 (SV40) staining

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enver Akalin, MD, Principal Investigator — Montefiore Medical Center/AECOM
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Everolimus (Zortress)+ Mycophenolic Acid(Myfortic): Everolimus: Starting dose 1.5 mg bid, target trough level 6-10 ng/ml. Myfortic Min. dose 360 mg bid and Max dose 720 mg bid. Both for one year.
- Reduced Dose Prograf+ Mycophenolic Acid(Myfortic): Tacrolimus: Target trough level of Tacrolimus 3-5 ng/ml. Myfortic Min. 360 mg bid and Max. 720 mg bid Both for one year.
Period: Overall Study
Arm/Group | Everolimus (Zortress)+ Mycophenolic Acid(Myfortic) | Reduced Dose Prograf+ Mycophenolic Acid(Myfortic)
Started | 2 | 0
Completed | 0 | 0
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: We did not analyze the data due to no patient enrolled in reduced dose prograf group and 2 patients enrolled in everolimus group did not complete the study due to death and adverse event
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus (Zortress)+ Mycophenolic Acid(Myfortic) | Reduced Dose Prograf+ Mycophenolic Acid(Myfortic) | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (2) |  | 63 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  | 2
  Male | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 1 |  | 1
  White | 0 |  | 0
  More than one race | 1 |  | 1
  Unknown or Not Reported | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in eGFR (Creatinine Clearance) as Measured by Serum Creatinine Blood Test
Description: Estimated glomerular filtration rate (eGFR) indicates kidney function. Normal eGFR value for healthy is 80-120ml/min. For transplants, it is expected to be 60-80 ml/min.
Time Frame: Baseline, One year
Population: The only two patients enrolled did not reach the one year mark; they did not complete the study so there was no data to analyze.
Arm/Group | Everolimus (Zortress)+ Mycophenolic Acid(Myfortic) | Reduced Dose Prograf+ Mycophenolic Acid(Myfortic)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The only two patients enrolled in everolimus group did not complete the study due to events leading to death and one due to proteinuria. The first participant was enrolled in March of 2012 and the study was terminated in August 2012.
Description: The two patients enrolled in everolimus group did not complete the study due to events leading to death and one due to proteinuria discontinued everolimus and switched to tacrolimus. The death occurred two months after enrollment. The proteinuria event occurred fours months after enrollment. No patient enrolled in reduced tacrolimus dose group and due to difficulty in enrollment the study is terminated. No data was analyzed for any participant.
Arm/Group | Everolimus (Zortress)+ Mycophenolic Acid(Myfortic) | Reduced Dose Prograf+ Mycophenolic Acid(Myfortic)
All-Cause Mortality (participants affected / at risk) | 1/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everolimus (Zortress)+ Mycophenolic Acid(Myfortic) (N=2) | Reduced Dose Prograf+ Mycophenolic Acid(Myfortic) (N=0)
proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) — proteinuria
Small bowel obstruction leading to death (Gastrointestinal disorders) | 1 (1) | 0 (0) — Small bowel obstruction lead to sepsis which lead to death

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No